CLINICAL TRIAL: NCT03989531
Title: Investigator-initiated, Placebo-controlled, Double-blind, Multi-center, Randomized Trial to Assess the Efficacy and Safety of Adrecizumab in Subjects With Cardiogenic Shock
Brief Title: Adrecizumab in Cardiogenic Shock
Acronym: ACCOST-HH
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dr. med. Mahir Karakas (Other)
Responsible Party: Sponsor-Investigator, Dr. med. Mahir Karakas, PD Dr Mahir Karakas, MBA, Universitätsklinikum Hamburg-Eppendorf
Organization: Universitätsklinikum Hamburg-Eppendorf (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Accost
Record Dates: First submitted 2019-06-17; First posted 2019-06-18 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-10

CONDITIONS: Cardiogenic Shock; Endothelial Dysfunction
Keywords: Cardiogenic Shock; Adrecizumab; Vascular integrity; Endothelial dysfunction
MeSH Terms: conditions — Shock, Cardiogenic | interventions — enibarcimab; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Adrecizumab on top of standard of care (Experimental): 8 mg/kg body weight Adrecizumab diluted in up to 100 mL saline as single dose infusion
  Interventions: Biological: Adrecizumab
- Placebo on top of standard of care (Placebo Comparator): 100 mL saline as single dose infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Adrecizumab — Drip infusion over 60 minutes
  Arms: Adrecizumab on top of standard of care
Drug: Placebo — Drip infusion over 60 minutes
  Other Names: Saline
  Arms: Placebo on top of standard of care

SUMMARY:
Cardiogenic shock is a serious medical condition with high mortality and morbidity. This trial assesses safety, tolerability and efficacy of Adrecizumab on top of standard of care in patients with cardiogenic shock.

DETAILED DESCRIPTION:
Despite optimal treatment the mortality in patients with cardiogenic shock still exceeds 50% and surviving patients mostly suffer from severe heart failure due to an impaired cardiac function.It is hypothesized, that Adrenomedullin is a key player in the (dys)-regulation of vascular integrity. Adrecizumab is the first-in-class humanized monoclonal anti-Adrenomedullin antibody, and acts as a long-lasting plasma Adrenomedullin enhancer stabilizing barrier function at a reasonable safety profile.When the anti-Adrenomedullin antibody Adrecizumab is administered in the blood circulation at high concentrations by far exceeding those of plasma Adrenomedullin, the compartmental distribution of Adrenomedullin is altered. Adrecizumab, an IgG with a molecular weight of more than 150 kDa, is too large to freely diffuse from the blood circulation to the interstitium. With its fast association kinetics Adrecizumab quickly binds to Adrenomedullin in the blood circulation and "pulls" Adrenomedullin, which has been initially located in the interstitium, from this compartment to the blood circulation. The more Adrecizumab is applied, the stronger is the "pulling" effect and the higher the resulting concentrations of Adrecizumab-bound Adrenomedullin in the blood circulation. The increase of Adrecizumab-bound Adrenomedullin in the blood circulation occurs within 5-15 minutes after administration of Adrecizumab, since it induces a translocation of preformed Adrenomedullin. As a consequence of this redistribution, the Adrenomedullin concentration in the interstitium decreases, and less Adrenomedullin is able to act on smooth muscle cells to exert its vasodilatative activity. In the progression to cardiogenic shock, when it comes to excessive vasodilation and hypotension, administration of Adrecizumab thus can reduce vasodilation by substracting excessive levels of interstitially located Adrenomedullin.

ELIGIBILITY:
Inclusion Criteria:

-Hospitalization for Cardiogenic shock (at the discretion of the local investigator)

Cardiogenic shock is usually defined as:

* Systolic blood pressure < 90 mmHg > 30 min or inotropes required to maintain pressure > 90 mmHg during systole
* Signs of left heart insufficiency and/ or pulmonary congestion
* Signs of impaired organ perfusion with at least one of the following:
* Altered mental status
* Cold, clammy skin
* Urine output <30 ml/h
* Serum lactate >2mmol/l

  * Age above 18 years at time of screening
  * Body weight below 150 kg at time of screening
  * Females/Males who agree to comply with the applicable contraceptive requirements of the protocol

Exclusion Criteria:

* Cardiogenic shock due to significant arrhythmias, which include any of the following: sustained ventricular tachycardia, bradycardia with sustained ventricular rate <35 beats per minute, or atrial fibrillation/ flutter with sustained ventricular response of >160 beats per minute
* Cardiogenic shock due to left ventricular outflow obstruction, obstructive hypertrophic cardiomyopathy or severe aortic stenosis (i.e., aortic valve area <0.8 cm2 or mean gradient >50 mmHg on prior or current echocardiogram), and severe mitral stenosis
* Cardiogenic shock due to mechanical cause or severe bleeding
* Cardiogenic shock due to untreated clinically significant CAD requiring revascularization
* Resuscitation > 60 minutes
* Severe pre-existing hepatic disease unrelated to cardiogenic shock
* Severe pre-existing renal disease (dialysis) unrelated to cardiogenic shock etiology

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2021-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Need of cardiovascular organ support within the first 30 days | 30 days
  Number of days through day 30 without need for cardiovascular organ support, including vasopressors, or mechanical support (VA-ECMO, Impella)

SECONDARY OUTCOMES:
30-day-Mortality | 30 days
  All-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mahir Karakas, MD, MBA, Principal Investigator — University Heart Center Hamburg
Locations (3):
- Germany (3):
  - University of Berlin, Campus Benjamin-Franklin, Berlin
  - University Heart Center Hamburg, Hamburg
  - University of Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karakas M, Akin I, Burdelski C, Clemmensen P, Grahn H, Jarczak D, Kessler M, Kirchhof P, Landmesser U, Lezius S, Lindner D, Mebazaa A, Nierhaus A, Ocak A, Rottbauer W, Sinning C, Skurk C, Soffker G, Westermann D, Zapf A, Zengin E, Zeller T, Kluge S. Single-dose of adrecizumab versus placebo in acute cardiogenic shock (ACCOST-HH): an investigator-initiated, randomised, double-blinded, placebo-controlled, multicentre trial. Lancet Respir Med. 2022 Mar;10(3):247-254. doi: 10.1016/S2213-2600(21)00439-2. Epub 2021 Dec 8. PMID 34895483